CLINICAL TRIAL: NCT02499536
Title: Relationship Between Intraoperative Atelectasis Findings on Transthoracic Lung Ultrasound and PaO2/FiO2
Brief Title: Relationship Between Atelectasis on Ultrasound and PaO2/FiO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Dr. Koh, Jae Chul, MD, Department of anesthesiology and pain medicine, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0189-002
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Atelectasis, Postoperative
Keywords: Atelectasis; Postoperative; Lung ultrasound
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study participants (Experimental): After general anesthesia development of the atelectasis will be investigated by the lung ultrasound
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Juxtapleural consolidation, loss of A lines, presence of B lines, air bronchogram, loss of sliding sign and presence of pulse sign on lung ultrasound finding will be investigated and recorded.

SUMMARY:
The aim of this study is to find out relationship between PaO2/FiO2 and atelectasis finding on intraoperative lung ultrasound.

DETAILED DESCRIPTION:
Patients aged 20~65 with ASA class (American Society of Anesthesiologists physical status classification) 1 or 2 who are scheduled to undergo general anesthesia by using endotracheal intubation and arterial line cannulation will participate in this study. The patients with abnormal chest x-ray finding, pregnancy, arrhythmia, ischemic heart disease will be excluded from this study as well as the patients who are scheduled to undergo lung or heart surgery.

After 5 minutes preoxygenation, patients will be monitored with pulse oxymetry, noninvasive blood pressure. General anesthesia will be proceeded with typical method and endotracheal intubation and arterial cannulation will be proceeded. After ventilator adjustment (tidal volume as 8 times of the patient's ideal body weight), airway pressures(peak and plateau) will be recorded. Subsequently, arterial blood sampling will be proceeded while examination of the atelectasis findings on lung ultrasound before surgery. Lung ultrasound examination will be proceeded on 6 sections of patient's basal segments of the lung, including anterior, lateral, posterior segment. Juxtapleural consolidation, loss of A lines, presence of B lines, air bronchogram, loss of sliding sign and presence of pulse sign on lung ultrasound finding will be investigated and recorded.

Same ultrasound examination and arterial blood sampling will be followed after surgery ends.

The results of PaO2/FiO2 on arterial blood samplings will be compared with findings on lung ultrasound before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20~65
* with ASA class 1 or 2
* who are scheduled to undergo general anesthesia by using endotracheal intubation and arterial line cannulation

Exclusion Criteria:

* The patients with abnormal chest x-ray finding,
* pregnancy,
* arrhythmia,
* ischemic heart disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Intraoperative lung ultrasound for atelectasis | Baseline (Before surgery begins) and Postoperative (Just after the surgery ends)
  Lung ultrasound examination for atelectasis findings (eg. whether there is a loss of A line or presence of B lines before and after surgery)
Change in PaO2/FiO2 | Baseline (Before surgery begins) and Postoperative (Just after the surgery ends)
  Arterial blood sampling to find out whether their is a change in PaO2/FiO2 before and after surgery.

SECONDARY OUTCOMES:
Airway pressure change | Baseline (Before surgery begins) and Postoperative (Just after the surgery ends)
  To find out if there is any difference between preoperative and postoperative airway pressures(peak and plateau pressure), monitored by ventilator used during general anesthesia in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ji young Kim, MD, PhD, Study Director — Department of anesthesiology and pain medicine, Gangnam Severance hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, Gangnam-gu, South Korea

REFERENCES:
- [Background] Lichtenstein D, Meziere G, Seitz J. The dynamic air bronchogram. A lung ultrasound sign of alveolar consolidation ruling out atelectasis. Chest. 2009 Jun;135(6):1421-1425. doi: 10.1378/chest.08-2281. Epub 2009 Feb 18. PMID 19225063